CLINICAL TRIAL: NCT05159141
Title: The Role of Circadian Rhythm in the Effect of Sleep Intervention on Obesity Prevention in Early Childhood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Sijia Gu, staff of Research Department, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCMCIRB-Y2020006
Record Dates: First submitted 2021-04-01; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Infant Sleep Problem
Keywords: Sleep; Obesity prevention; Circadian rhythm; Children; Behavioral intervention

STUDY DESIGN:
Intervention Model Description: Infants are randomly assigned to one of two groups: Behavioral Sleep Intervention or Control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Trial participants and individuals assessing the outcomes are blinded to the participant's condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Infant sleep monitoring (Actigraphy and sleep dairy) and parental surveys
- Infant behavioral sleep intervention (Experimental): Interventionists collaborate with the family to design a tailored sleep intervention strategy, which involves appropriate sleep schedule and bedtime routine, putting the child to bed while still sleepy rather than when already asleep, and waiting 1 to 2 minutes before attending to the child during nocturnal awakenings. Parents are educated to implement the behavioral protocol at bedtime and subsequent night wakings.
  Interventions: Behavioral: Behavioral sleep intervention

INTERVENTIONS:
Behavioral: Behavioral sleep intervention — The intervention consists of an infant behavioral sleep protocol. In the tailored intervention approach, parents are asked to implement the behavioral protocol at bedtime and at subsequent night wakings.
  Arms: Infant behavioral sleep intervention

SUMMARY:
Over the last 40 years, obesity has increased dramatically among all age groups, especially in infants and young children, and became an important global public health challenge, thus early prevention is the highest priority. Emerging studies have found that infant sleep intervention is very likely to become one of the most important strategies for early obesity prevention. However, its action path is not clear, making the target of sleep intervention relatively vague. The role of circadian rhythm in human health status has received increasing attention in recent years. Both animal experiment-based studies and adult clinic-based studies have found significant effect of the circadian rhythm on obesity and other metabolic disorders. Therefore, the present research will establish a community-based 1:1 parallel multi-center randomized controlled trial of sleep intervention cohort in communities with highly rapid weight gain at the early infancy stage. Investigators will collect daily rhythm data, including sleep-wake rhythm, rest-activity rhythm, light-dark cycle, and feeding-fasting, as well as the real-world golden standard of circadian rhythm assessed by seven times saliva melatonin, to test the impact of the sleep intervention program, to determine the causal mechanism of circadian rhythm in the occurrence&nbsp;and&nbsp; development of obesity and metabolic disorder early in life. Our study will provide a new theoretical basis for the establishment of the stable circadian rhythm for the prevention of infant obesity, which has important public health significance.

DETAILED DESCRIPTION:
1. Research content 1.1 Study on the Reliability and Validity of Daily Circadian Rhythm of Infant and Young Child Behavior and Establishment of Circadian Circadian Rhythm Prediction Model In three study communities, 10 infants aged 4 months, 6 months, 12 months and 2 years old were recruited, with a total of 120 infants. Daily rhythms of sleep, activity, illumination and eating were collected by using portable device Actiwatch-2 and daily log book. Saliva at 7 time points (09: 00, 13: 00, 17: 00, 21: 00, 01: 00, 05: 00 and 09: 00) were collected to determine the level of melatonin as the gold standard for circadian rhythm of biological clocks under natural environment. The correlation between daily circadian rhythms and characteristics of melatonin secretion was determined. A model with high reliability was established by mathematical modeling.

   1.2 Multicenter Cohort Study of Effects of Sleep Intervention on Metabolic Function in Childhood Obesity Methods: A 1: 1 parallel multicenter randomized controlled trial was conducted to recruit 80 infants from each of the control group and the intervention group at 28 days after birth. The control group was followed up for 5 times (28 days, 2 months, 4 months, 6 months and 12 months) of evidence-based infant sleep intervention on the basis of routine child care, and followed up until 2 years old. The main outcomes were changes in BMI z at 0-6 months of age and metabolic markers of obesity at 2 years of age, such as BMI z, subcutaneous fat, body composition and blood biochemistry. On the basis of descriptive analysis, the effects of sleep intervention on infant obesity metabolism and daily rhythm were determined, and the causal mechanism of circadian rhythm, obesity metabolic index and other factors were determined by using Bayesian causal network.

   1.3 Verification of Predictive Models for Circadian Rhythms of Behavioral Clocks In the second part of the three study communities, the two groups were randomly selected 20 cases, a total of 120 infants and children.

   At 4 months, 6 months, 12 months and 2 years of age after birth, saliva samples were collected at 2 time points in addition to Actiwatch-2 and daily rhythm data, and melatonin levels were measured to validate the rhythm prediction model.
2. Research objectives

Based on the concept of early prevention, this project focuses on the role of circadian rhythms in infant sleep intervention to prevent obesity and accomplishes the following two objectives:

2.1 To determine the intensity of correlation between the daily rhythm of infants and the characteristics of melatonin secretion rhythm of gold standard.

Over mathematical modeling to establish high reliability and validity of behavioral biological clock circadian rhythm prediction model in infants and young children to verify and apply to sleep intervention multicenter cohort study.

2.2 To explore the effect of sleep intervention on infants by establishing a standard multicenter cohort of infant sleep intervention It is of great public health significance to provide high quality evidence for early prevention and control of childhood obesity and to design more pertinent prevention and control strategies.

ELIGIBILITY:
Inclusion Criteria:

* Infants and young children: age 4 months, 6 months, 12 months, and 2 years old;
* term single birth (37-42 weeks of gestation);
* health inactive disease;
* normal Griffiths developmental assessment;
* natural vaginal delivery or social cesarean section;
* Apgar score greater than 7 at birth for 1 or 5 minute.

Exclusion Criteria:

* Infants and young children: birth weight < 2500 g;
* premature or multiple births;
* prenatal ultrasonography indicating intrauterine growth retardation;
* severe organic diseases of the baby after birth that have been hospitalized for treatment;
* congenital malformations or diseases affecting the feeding of the baby (cleft lip and palate, metabolic diseases, etc.).

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Children's sleep condition | 4 months old
  A 7-day assessment of children's sleep condition was conducted by using Actiwatch (AMI) and a sleep diary. AMI is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children's sleep condition | 6 months old
  A 7-day assessment of children's sleep condition was conducted by using Actiwatch (AMI) and a sleep diary. AMI is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children's sleep condition | 12 months old
  A 7-day assessment of children's sleep condition was conducted by using Actiwatch (AMI) and a sleep diary. AMI is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children's sleep condition | 2 years old
  A 7-day assessment of children's sleep condition was conducted by using Actiwatch (AMI) and a sleep diary. AMI is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children's anthropometrics | 4 months old
  Weight in kilograms
Children's anthropometrics | 6 months old
  Weight in kilograms
Children's anthropometrics | 12 months old
  Weight in kilograms
Children's anthropometrics | 2 years old
  Weight in kilograms
Children's anthropometrics | 4 months old
  Length/height in centimeters
Children's anthropometrics | 6 months old
  Length/height in centimeters
Children's anthropometrics | 12 months old
  Length/height in centimeters
Children's anthropometrics | 2 years old
  Length/height in centimeters
Children's anthropometrics | 4 months old
  Weight and height will be combined to report BMI (calculated by weight divided by the square of length/height) in kg/m^2
Children's anthropometrics | 6 months old
  Weight and height will be combined to report BMI (calculated by weight divided by the square of length/height) in kg/m^2
Children's anthropometrics | 12 months old
  Weight and height will be combined to report BMI (calculated by weight divided by the square of length/height) in kg/m^2
Children's anthropometrics | 2 years old
  Weight and height will be combined to report BMI (calculated by weight divided by the square of length/height) in kg/m^2
Children's anthropometrics | 6 months old
  Arm circumference in centimeters
Children's anthropometrics | 12 months old
  Arm circumference in centimeters
Children's anthropometrics | 2 years old
  Arm circumference in centimeters
Children's anthropometrics | 6 months old
  Triceps skinfold thicknesses in centimeters
Children's anthropometrics | 12 months old
  Triceps skinfold thicknesses in centimeters
Children's anthropometrics | 2 years old
  Triceps skinfold thicknesses in centimeters
Children's anthropometrics | 6 months old
  Subscapular skinfold thicknesses in centimeters
Children's anthropometrics | 12 months old
  Subscapular skinfold thicknesses in centimeters
Children's anthropometrics | 2 years old
  Subscapular skinfold thicknesses in centimeters
Infant metabolism index | 2 years old
  Blood total cholesterol level
Infant metabolism index | 2 years old
  Blood high-density lipoprotein level
Infant metabolism index | 2 years old
  Blood low-density lipoprotein level
Infant metabolism index | 2 years old
  Blood triglycerides level
Infant metabolism index | 2 years old
  Fasting blood glucose level
Infant metabolism index | 2 years old
  Blood insulin level
Infant metabolism index | 2 years old
  Blood ghrelin level
Infant metabolism index | 2 years old
  Blood leptin level
Infant metabolism index | 2 years old
  Blood adiponectin level
Children's circadian rhythm | 4 months old
  Saliva melatonin levels at 7 Time Points (09: 00, 13: 00, 17: 00, 21: 00, 01: 00, 05: 00 and 09: 00) as the gold standard for circadian rhythms of biological clocks under natural environment.
Children's circadian rhythm | 6 months old
  Saliva melatonin levels at 7 Time Points (09: 00, 13: 00, 17: 00, 21: 00, 01: 00, 05: 00 and 09: 00) as the gold standard for circadian rhythms of biological clocks under natural environment.
Children's circadian rhythm | 12 months old
  Saliva melatonin levels at 7 Time Points (09: 00, 13: 00, 17: 00, 21: 00, 01: 00, 05: 00 and 09: 00) as the gold standard for circadian rhythms of biological clocks under natural environment.
Children's circadian rhythm | 2 years old
  Saliva melatonin levels at 7 Time Points (09: 00, 13: 00, 17: 00, 21: 00, 01: 00, 05: 00 and 09: 00) as the gold standard for circadian rhythms of biological clocks under natural environment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Fan, PhD, Study Chair — Shanghai children's medicial center affiliated shanghai jiaotong University School of Medicine
Locations (1):
- Shanghai children's medicial center affiliated shanghai jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
not yet decided

REFERENCES:
- [Background] Komarzynski S, Bolborea M, Huang Q, Finkenstadt B, Levi F. Predictability of individual circadian phase during daily routine for medical applications of circadian clocks. JCI Insight. 2019 Sep 19;4(18):e130423. doi: 10.1172/jci.insight.130423. PMID 31430260
- [Result] WHO-UNICEF- Lancet Commissioners. After COVID-19, a future for the world's children? Lancet. 2020 Aug 1;396(10247):298-300. doi: 10.1016/S0140-6736(20)31481-1. Epub 2020 Jul 2. No abstract available. PMID 32622373
- [Result] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Result] Sung H, Siegel RL, Torre LA, Pearson-Stuttard J, Islami F, Fedewa SA, Goding Sauer A, Shuval K, Gapstur SM, Jacobs EJ, Giovannucci EL, Jemal A. Global patterns in excess body weight and the associated cancer burden. CA Cancer J Clin. 2019 Mar;69(2):88-112. doi: 10.3322/caac.21499. Epub 2018 Dec 12. PMID 30548482
- [Result] Geserick M, Vogel M, Gausche R, Lipek T, Spielau U, Keller E, Pfaffle R, Kiess W, Korner A. Acceleration of BMI in Early Childhood and Risk of Sustained Obesity. N Engl J Med. 2018 Oct 4;379(14):1303-1312. doi: 10.1056/NEJMoa1803527. PMID 30281992
- [Result] Ward ZJ, Long MW, Resch SC, Giles CM, Cradock AL, Gortmaker SL. Simulation of Growth Trajectories of Childhood Obesity into Adulthood. N Engl J Med. 2017 Nov 30;377(22):2145-2153. doi: 10.1056/NEJMoa1703860. PMID 29171811
- [Result] Juonala M, Magnussen CG, Berenson GS, Venn A, Burns TL, Sabin MA, Srinivasan SR, Daniels SR, Davis PH, Chen W, Sun C, Cheung M, Viikari JS, Dwyer T, Raitakari OT. Childhood adiposity, adult adiposity, and cardiovascular risk factors. N Engl J Med. 2011 Nov 17;365(20):1876-85. doi: 10.1056/NEJMoa1010112. PMID 22087679
- [Result] Franks PW, Hanson RL, Knowler WC, Sievers ML, Bennett PH, Looker HC. Childhood obesity, other cardiovascular risk factors, and premature death. N Engl J Med. 2010 Feb 11;362(6):485-93. doi: 10.1056/NEJMoa0904130. PMID 20147714
- [Result] Fontaine KR, Redden DT, Wang C, Westfall AO, Allison DB. Years of life lost due to obesity. JAMA. 2003 Jan 8;289(2):187-93. doi: 10.1001/jama.289.2.187. PMID 12517229
- [Result] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Result] Hamilton D, Dee A, Perry IJ. The lifetime costs of overweight and obesity in childhood and adolescence: a systematic review. Obes Rev. 2018 Apr;19(4):452-463. doi: 10.1111/obr.12649. Epub 2017 Dec 22. PMID 29271111
- [Result] Sonntag D, Ali S, De Bock F. Lifetime indirect cost of childhood overweight and obesity: A decision analytic model. Obesity (Silver Spring). 2016 Jan;24(1):200-6. doi: 10.1002/oby.21323. Epub 2015 Dec 6. PMID 26638187
- [Result] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Result] Hale L, Troxel W, Buysse DJ. Sleep Health: An Opportunity for Public Health to Address Health Equity. Annu Rev Public Health. 2020 Apr 2;41:81-99. doi: 10.1146/annurev-publhealth-040119-094412. Epub 2020 Jan 3. PMID 31900098
- [Result] Zhu B, Shi C, Park CG, Zhao X, Reutrakul S. Effects of sleep restriction on metabolism-related parameters in healthy adults: A comprehensive review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2019 Jun;45:18-30. doi: 10.1016/j.smrv.2019.02.002. Epub 2019 Feb 10. PMID 30870662
- [Result] Piovezan RD, Hirotsu C, Moizinho R, de Sa Souza H, D'Almeida V, Tufik S, Poyares D. Associations between sleep conditions and body composition states: results of the EPISONO study. J Cachexia Sarcopenia Muscle. 2019 Oct;10(5):962-973. doi: 10.1002/jcsm.12445. Epub 2019 May 24. PMID 31125517
- [Result] Jiang F, Zhu S, Yan C, Jin X, Bandla H, Shen X. Sleep and obesity in preschool children. J Pediatr. 2009 Jun;154(6):814-8. doi: 10.1016/j.jpeds.2008.12.043. Epub 2009 Feb 24. PMID 19243786
- [Result] Jiang YR, Spruyt K, Chen WJ, Shen XM, Jiang F. Somatic growth of lean children: the potential role of sleep. World J Pediatr. 2014 Aug;10(3):245-50. doi: 10.1007/s12519-014-0500-2. Epub 2014 Aug 15. PMID 25124976
- [Result] Jiang YR, Spruyt K, Chen WJ, Mei H, Sun WQ, Wang Y, Li SH, Luo ZC, Shen XM, Jiang F. Associations between parent-reported sleep duration and adiposity in Chinese early adolescents. J Public Health (Oxf). 2015 Jun;37(2):277-85. doi: 10.1093/pubmed/fdu049. Epub 2014 Aug 7. PMID 25104839
- [Result] Deng Y, Wang G, Ye X, Jiang Y, Lin Q, Dong S, Song Y, Zhu L, Meng M, Li W, Zhu Q, Sun W, Jiang F. The association between 25-hydroxyvitamin D levels and children's sleep-wake patterns: a prospective cohort study. Sleep Med. 2020 Mar;67:207-214. doi: 10.1016/j.sleep.2019.11.1252. Epub 2019 Dec 12. PMID 31952028
- [Result] Paul IM, Savage JS, Anzman-Frasca S, Marini ME, Beiler JS, Hess LB, Loken E, Birch LL. Effect of a Responsive Parenting Educational Intervention on Childhood Weight Outcomes at 3 Years of Age: The INSIGHT Randomized Clinical Trial. JAMA. 2018 Aug 7;320(5):461-468. doi: 10.1001/jama.2018.9432. PMID 30088009
- [Result] Savage JS, Birch LL, Marini M, Anzman-Frasca S, Paul IM. Effect of the INSIGHT Responsive Parenting Intervention on Rapid Infant Weight Gain and Overweight Status at Age 1 Year: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):742-9. doi: 10.1001/jamapediatrics.2016.0445. PMID 27271455
- [Result] Taylor RW, Gray AR, Heath AM, Galland BC, Lawrence J, Sayers R, Healey D, Tannock GW, Meredith-Jones KA, Hanna M, Hatch B, Taylor BJ. Sleep, nutrition, and physical activity interventions to prevent obesity in infancy: follow-up of the Prevention of Overweight in Infancy (POI) randomized controlled trial at ages 3.5 and 5 y. Am J Clin Nutr. 2018 Aug 1;108(2):228-236. doi: 10.1093/ajcn/nqy090. PMID 30101329
- [Result] Taylor BJ, Gray AR, Galland BC, Heath AM, Lawrence J, Sayers RM, Cameron S, Hanna M, Dale K, Coppell KJ, Taylor RW. Targeting Sleep, Food, and Activity in Infants for Obesity Prevention: An RCT. Pediatrics. 2017 Mar;139(3):e20162037. doi: 10.1542/peds.2016-2037. PMID 28242860
- [Result] Hernandez-Garcia J, Navas-Carrillo D, Orenes-Pinero E. Alterations of circadian rhythms and their impact on obesity, metabolic syndrome and cardiovascular diseases. Crit Rev Food Sci Nutr. 2020;60(6):1038-1047. doi: 10.1080/10408398.2018.1556579. Epub 2019 Jan 11. PMID 30633544
- [Result] Albrecht U, Ripperger JA. Circadian Clocks and Sleep: Impact of Rhythmic Metabolism and Waste Clearance on the Brain. Trends Neurosci. 2018 Oct;41(10):677-688. doi: 10.1016/j.tins.2018.07.007. Epub 2018 Sep 25. PMID 30274603
- [Result] Kuhlman SJ, Craig LM, Duffy JF. Introduction to Chronobiology. Cold Spring Harb Perspect Biol. 2018 Sep 4;10(9):a033613. doi: 10.1101/cshperspect.a033613. PMID 29038118
- [Result] Lewis P, Foster RG, Erren TC. Ticking time bomb? High time for chronobiological research. EMBO Rep. 2018 May;19(5):e46073. doi: 10.15252/embr.201846073. Epub 2018 Apr 3. PMID 29615393
- [Result] Panda S. The arrival of circadian medicine. Nat Rev Endocrinol. 2019 Feb;15(2):67-69. doi: 10.1038/s41574-018-0142-x. No abstract available. PMID 30602736
- [Result] Burki T. Nobel Prize awarded for discoveries in circadian rhythm. Lancet. 2017 Oct 14;390(10104):e25. doi: 10.1016/S0140-6736(17)32661-2. Epub 2017 Oct 12. No abstract available. PMID 29047447
- [Result] Mohawk JA, Green CB, Takahashi JS. Central and peripheral circadian clocks in mammals. Annu Rev Neurosci. 2012;35:445-62. doi: 10.1146/annurev-neuro-060909-153128. Epub 2012 Apr 5. PMID 22483041
- [Result] Flanagan A, Bechtold DA, Pot GK, Johnston JD. Chrono-nutrition: From molecular and neuronal mechanisms to human epidemiology and timed feeding patterns. J Neurochem. 2021 Apr;157(1):53-72. doi: 10.1111/jnc.15246. Epub 2020 Dec 10. PMID 33222161
- [Result] Mason IC, Qian J, Adler GK, Scheer FAJL. Impact of circadian disruption on glucose metabolism: implications for type 2 diabetes. Diabetologia. 2020 Mar;63(3):462-472. doi: 10.1007/s00125-019-05059-6. Epub 2020 Jan 8. PMID 31915891
- [Result] Chellappa SL, Vujovic N, Williams JS, Scheer FAJL. Impact of Circadian Disruption on Cardiovascular Function and Disease. Trends Endocrinol Metab. 2019 Oct;30(10):767-779. doi: 10.1016/j.tem.2019.07.008. Epub 2019 Aug 16. PMID 31427142
- [Result] Rust MJ, Golden SS, O'Shea EK. Light-driven changes in energy metabolism directly entrain the cyanobacterial circadian oscillator. Science. 2011 Jan 14;331(6014):220-3. doi: 10.1126/science.1197243. PMID 21233390
- [Result] Turek FW, Joshu C, Kohsaka A, Lin E, Ivanova G, McDearmon E, Laposky A, Losee-Olson S, Easton A, Jensen DR, Eckel RH, Takahashi JS, Bass J. Obesity and metabolic syndrome in circadian Clock mutant mice. Science. 2005 May 13;308(5724):1043-5. doi: 10.1126/science.1108750. Epub 2005 Apr 21. PMID 15845877
- [Result] Jones ME, Schoemaker MJ, McFadden EC, Wright LB, Johns LE, Swerdlow AJ. Night shift work and risk of breast cancer in women: the Generations Study cohort. Br J Cancer. 2019 Jul;121(2):172-179. doi: 10.1038/s41416-019-0485-7. Epub 2019 May 29. PMID 31138896
- [Result] Vetter C, Dashti HS, Lane JM, Anderson SG, Schernhammer ES, Rutter MK, Saxena R, Scheer FAJL. Night Shift Work, Genetic Risk, and Type 2 Diabetes in the UK Biobank. Diabetes Care. 2018 Apr;41(4):762-769. doi: 10.2337/dc17-1933. Epub 2018 Feb 12. PMID 29440150
- [Result] Lin QM, Spruyt K, Leng Y, Jiang YR, Wang GH, Dong SM, Mei H, Jiang F. Cross-cultural disparities of subjective sleep parameters and their age-related trends over the first three years of human life: A systematic review and meta-analysis. Sleep Med Rev. 2019 Dec;48:101203. doi: 10.1016/j.smrv.2019.07.006. Epub 2019 Aug 5. PMID 31494051
- [Result] Ray S, Reddy AB. Cross-talk between circadian clocks, sleep-wake cycles, and metabolic networks: Dispelling the darkness. Bioessays. 2016 Apr;38(4):394-405. doi: 10.1002/bies.201500056. Epub 2016 Feb 11. PMID 26866932
- [Result] Goncalves BS, Adamowicz T, Louzada FM, Moreno CR, Araujo JF. A fresh look at the use of nonparametric analysis in actimetry. Sleep Med Rev. 2015 Apr;20:84-91. doi: 10.1016/j.smrv.2014.06.002. Epub 2014 Jun 20. PMID 25065908
- [Result] Yamazaki S, Kerbeshian MC, Hocker CG, Block GD, Menaker M. Rhythmic properties of the hamster suprachiasmatic nucleus in vivo. J Neurosci. 1998 Dec 15;18(24):10709-23. doi: 10.1523/JNEUROSCI.18-24-10709.1998. PMID 9852606
- [Result] Attanasio A, Borrelli P, Gupta D. Circadian rhythms in serum melatonin from infancy to adolescence. J Clin Endocrinol Metab. 1985 Aug;61(2):388-90. doi: 10.1210/jcem-61-2-388. PMID 4008613